CLINICAL TRIAL: NCT05373238
Title: Same Day Discharge After Laparoscopic Hysterectomy vs Late Discharge
Brief Title: Same Day Discharge After Laparoscopic Hysterectomy
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Caglar Cetin, Principal investigator, Bezmialem Vakif University
Other Study IDs: BVU-10.2021
Record Dates: First submitted 2022-05-05; First posted 2022-05-13 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Surgery--Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early Discharge: < discharge before 24 hours
  Interventions: Procedure: Early discharge
- Late Discharge: discharge after 24 hours
  Interventions: Procedure: Early discharge

INTERVENTIONS:
Procedure: Early discharge — Early discharge

SUMMARY:
Patients who are scheduled for laparoscopic hysterectomy will be included in the study.

After the operation, those who are well and without major distress will be discharged from the hospital before 24 hours. Those who have pain or have additional health problems will be observed further.

Our aim is to compare these two groups in terms of early complications and operation characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Patients Scheduled For Hysterectomy

Exclusion Criteria:

* Diagnosis of Malignancy
* Those with intraoperative complication

Ages: 35 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Female patients aged 35-80 scheduled for laparoscopic hysterectomy
Sampling Method: Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Complication in 30 days | 30 days
  Number of patients with surgical complications, postoperative complications, wound complications

SECONDARY OUTCOMES:
Postop hb | 30 day
  Number of patients whose hemoglobin value declined beyond two parameters. (mg/dL)
Postop htc | 30 day
  Number of patients whose hematocrit value declined more than 5 percent (%)

CONTACTS AND LOCATIONS:
Overall Officials: Gurkan Kiran, Study Chair — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided